CLINICAL TRIAL: NCT03393572
Title: Intraperitoneal Instillation of Bupivacaine With Either Magnesium Sulphate or Nalbuphine for Postoperative Pain Control in Laparoscopic Hysterectomy: a Prospective, Randomized, Double-blinded Trial.
Brief Title: Intraperitoneal Bupivacaine With Magnesium or Nalbuphine for Postoperative Pain Control in Laparoscopic Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Khairy Elbeialy, Lecturer of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU R49/2017
Record Dates: First submitted 2018-01-03; First posted 2018-01-08 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Anesthesia
MeSH Terms: interventions — Magnesium Sulfate; Nalbuphine; Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group BM (Active Comparator): bupivacaine 0.25% plus magnesium sulphate.
  Interventions: Drug: Bupivacaine 0.25%; Drug: Magnesium sulphate.
- Group BN (Active Comparator): bupivacaine 0.25% plus nalbuphine
  Interventions: Drug: Bupivacaine 0.25%; Drug: nalbuphine

INTERVENTIONS:
Drug: Bupivacaine 0.25% — Patients will receive 30 mL of intraperitoneal bupivacaine 0.25%
Drug: Magnesium sulphate. — Patients will receive intraperitoneal 30 mg/kg of magnesium sulphate.
  Arms: Group BM
Drug: nalbuphine — Patients will receive intraperitoneal 5 mg nalbuphine
  Other Names: opioid
  Arms: Group BN

SUMMARY:
The purpose of this study is to compare between the addition of Mg sulphate or Nalbuphine to intraperitoneal bupivacaine installation in laparoscopic hysterectomy for postoperative pain control and their relative adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I and II
* scheduled for laparoscopic hysterectomy

Exclusion Criteria:

* ASA physical status more than II
* Obesity (body mass index higher than 30 kg/ m2)
* History of chronic opioids intake
* Known hypomagnesaemia or hypermagnesaemia
* Chronic alcoholism
* Heart block
* Renal failure
* Patients with history of left ventricular failure
* Patients taking beta-blocking drugs
* Allergy to the study drugs
* if surgery changed to open hysterectomy,

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Rescue analgesia time | First 24 hours postoperatively
  Time to first analgesia requirment(considering the extubation is the zero time)

SECONDARY OUTCOMES:
Visual analogue scale [VAS] | First 24 hours postoperatively
  Visual analogue scale [VAS] will be used to measure pain score at 30 min, 1, 2, 4, 6, 8, 10, 12 and 24 h after surgery. All the study patients will be instructed about the use of the VAS scale before induction of anesthesia (VAS score 0 cm = no pain, VAS score 10 cm = worst possible pain)
Total analgesic consumption | First 24 hours postoperatively
  Intravenous diclofenac 75 mg will be given as rescue analgesic when VAS ≥ 4.Total diclofenac consumption will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Elbeialy, Cairo, Egypt